CLINICAL TRIAL: NCT06091436
Title: A Multicenter, Double-blind, Non-inferiority, Phase 3 RCT Comparing GenSci094 and Recombinant FSH During the First Seven Days of Ovarian Stimulation in Chinese ART Patients
Brief Title: To Investigate Efficacy and Safety of a Single Injection of GenSci094 for Ovarian Stimulation Using Daily Recombinant FSH as Reference
Acronym: ANGAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GenSci094-301
Record Dates: First submitted 2023-08-08; First posted 2023-10-19 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — follitropin alfa; ganirelix; Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GenSci094 (Experimental): Participants received a single subcutaneous (SC) injection of 150 µg or 100µg GenSci094 on day 2 or 3 of the menstrual cycle (Stimulation Day 1); 7 daily SC injections from Stimulation Days 1 to 7 with placebo-recFSH; followed by daily SC injections with 150 IU or225IU recFSH up to the day of hCG. Daily SC injections of Ganirelix were administered from Stimulation Day 5 to the day of hCG; at which time a single dose of hCG was given when 3 follicles >= 17 mm. On the day of oocyte pick up (OPU) daily doses of progesterone were started and continued for up to 6 weeks or menses.
  Interventions: Drug: GenSci094; Drug: Placebo RecFSH / follitropin alfa; Biological: RecFSH / Follitropin alfa (Days 8 to hCG); Drug: Ganirelix; Biological: hCG; Drug: Progesterone
- recFSH (Active Comparator): Participants received a single SC injection of placebo GenSci094 on day 2 or 3 of the menstrual cycle (Stimulation Day 1); 7 daily SC injections with 150 IU or 225IU recFSH from Stimulation Days 1 to 7; followed by daily SC injections with 200 IU recFSH up to the day of hCG. Daily SC injections of Ganirelix were given from Stimulation Day 5 to the day of hCG; at which time a single dose of hCG was administered when 3 follicles >= 17 mm. On the day of OPU daily doses of progesterone were started and continued for up to 6 weeks or menses.
  Interventions: Biological: Biological: RecFSH / Follitropin alfa (Days 1 to 7); Drug: Placebo GenSci094; Biological: RecFSH / Follitropin alfa (Days 8 to hCG); Drug: Ganirelix; Biological: hCG; Drug: Progesterone

INTERVENTIONS:
Drug: GenSci094 — On the morning of day 2 or 3 of the menstrual cycle (Stimulation Day 1), a single SC injection of 150 μg or 100μg (0.5 mL) GenSci094 was administered in the abdominal wall.
  Arms: GenSci094
Drug: Placebo RecFSH / follitropin alfa — powder-injection, but without the active ingedient, SC injection . Daily SC injections were started on Stimulation Day 1 and continued up to and including Stimulation Day 7.
  Arms: GenSci094
Biological: Biological: RecFSH / Follitropin alfa (Days 1 to 7) — Daily SC injections with 150IU or 225IU recFSH were started on Stimulation Day 1 and continued up to and including Stimulation Day 7.
  Arms: recFSH
Drug: Placebo GenSci094 — Pre-filled syringe containing an identical solution when compared to GenSci094. On the morning of day 2 or 3 of the menstrual cycle (Stimulation Day 1), a single SC injection was administered in the abdominal wall.
  Arms: recFSH
Biological: RecFSH / Follitropin alfa (Days 8 to hCG) — From Stimulation Day 8 onwards a daily SC dose 75IU～300 IU recFSH was administered up to and including the Day of hCG.
Drug: Ganirelix — On Stimulation Day 5 a daily SC injection of 0.25 mg was started, which continued up to and including the day of hCG
Biological: hCG — When 3 follicles >= 17 mm were observed by USS, a single dose of 10,000 IU/USP hCG was administered; or, for those at risk for Ovarian Hyperstimulation Syndrome (OHSS), a lower dose of 5,000 IU/USP
Drug: Progesterone — On the day of OPU, luteal phase support was started by administering micronized progesterone of at least 400 mg/day vaginally, and 40mg/d oral, which continued for at least 6 weeks, or up to menses.

SUMMARY:
To investigate the efficacy and safety of a single injection of GenSci094 to induce multi-follicular development for controlled ovarian stimulation using daily recombinant FSH (recFSH) as a reference. The primary hypothesis is that a single injection of GenSci094 is non-inferior to daily treatment with recFSH in initiating multi-follicular growth.

ELIGIBILITY:
Inclusion Criteria:

* Females of couples with an indication for Controlled Ovarian Stimulation (COS) and in-vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI);
* >=20 and <40 years of age at the time of signing informed consent;
* Body weight >=50 kg and body mass index (BMI) >=18 and <=28 kg/m^2;
* AMH<4.0 and>=1.1μg/L FSH<10 IU/L
* Willing and able to sign informed consent.

Exclusion Criteria:

* History of ovarian hyper-response or ovarian hyperstimulation syndrome (OHSS);
* History of/or current polycystic ovary syndrome (PCOS);
* More than 20 basal antral follicles <11 mm (both ovaries combined) as measured on ultrasound scan (USS) in the early follicular phase (menstrual cycle day 2-4);
* Presence of unilateral or bilateral hydrosalphinx (visible on USS);
* Presence of any clinically relevant pathology affecting the uterine cavity or fibroids >4 cm;
* More than three unsuccessful IVF cycles since the last established ongoing pregnancy (if applicable);
* History of non- or low ovarian response to FSH/ human menopausal gonadotropin (hMG) treatment;
* History of recurrent miscarriage (3 or more, even when unexplained);
* Any clinically relevant abnormal laboratory value based on a sample taken during the screening phase;
* Contraindications for the use of gonadotropins (e.g. tumors, pregnancy/lactation, undiagnosed vaginal bleeding, hypersensitivity, ovarian cysts);
* Recent history of/or current epilepsy, human immunodeficiency virus (HIV) infection, diabetes, cardiovascular, gastro-intestinal, hepatic, renal or pulmonary disease;
* Use of hormonal preparations within 1 month prior to randomization;
* Hypersensitivity to any of the concomitant medication prescribed as part of the treatment regimen in this protocol;
* Administration of investigational drugs within three months prior to signing informed consent.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Mean Number of Oocytes Retrieved | Approximately Day 10-14

SECONDARY OUTCOMES:
Percentage of Participants With an Ongoing Pregnancy (Ongoing Pregnancy Rate) | Assessed at least 10 weeks after embryo transfer
Percentage of Fertilized Oocytes (Fertilization Rate) | Up to 18 hours after start of fertilization
Number of Embryos Obtained on Day 3 Categorized by Quality | Post fertilization Day 3
Percentage of Gestational Sacs (Implantation Rate) | Up to 6 weeks after embryo transfer
Percentage of Participants With a Biochemical Pregnancy Per Embryo Transfer | Two weeks after embryo transfe
Percentage of Participants With a early miscarriage（early miscarriage rate）Per Clinical Pregnancy | Up to 12 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: xiaoyan liang, doctor, Study Chair — The Sixth Affiliated Hospital, Sun Yat-sen University Guangdong Gastrointestinal Hospital
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University Guangdong Gastrointestinal Hospital, Guangzhou, Guangdong, China